CLINICAL TRIAL: NCT03425500
Title: Bridging Reconstruction of Massive Rotator Cuff Tears by Human Dermal Allograft Augmentation Compared to Superior Capsular Reconstruction
Brief Title: Massive Rotator Cuff Tear Reconstruction
Acronym: SCR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Ivan Wong, Orthopaedic Surgeon MD FRCS(C), Dip. Sports Medicine, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IW-002
Record Dates: First submitted 2018-01-31; First posted 2018-02-07 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Rotator Cuff Tear Arthropathy
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bridging Rotator Cuff Group (Experimental): Bridging Rotator Cuff Reconstruction of massive rotator cuff tear using GRAFTJACKET™ allograft.
  Interventions: Procedure: Bridging Rotator Cuff Reconstruction; Device: GRAFTJACKET™ allograft
- Superior Capsular Group (Active Comparator): Superior Capsular Reconstruction of massive rotator cuff tear
  Interventions: Procedure: Superior Capsular Reconstruction

INTERVENTIONS:
Procedure: Bridging Rotator Cuff Reconstruction — Bridging Rotator Cuff Reconstruction of massive rotator cuff tear using a GRAFTJACKET™ allograft
  Arms: Bridging Rotator Cuff Group
Procedure: Superior Capsular Reconstruction — Superior Capsular Reconstruction of massive rotator cuff tear
  Arms: Superior Capsular Group
Device: GRAFTJACKET™ allograft — The acellular human dermal allograft in used in the bridging rotator cuff reconstruction
  Other Names: Acellular human dermal allograft
  Arms: Bridging Rotator Cuff Group

SUMMARY:
To compare bridging reconstruction to superior capsular reconstruction using human dermal allograft augmentation for repair of massive rotator cuff tears.

DETAILED DESCRIPTION:
A total of 60 patients will be enrolled in the study. In the pre-operative period, there will be no additional time requirements for the patient, except for the informed consent process for the study. Routine radiographs including an AP and Y view of the shoulder as well as a pre-operative MRI are obtained for all patients undergoing rotator cuff surgery.

The patients will complete a structured clinical examination conducted by a sports medicine fellowship trained orthopaedic consultant. The examination will consist of range of motion testing by goniometer as well as strength testing by hand dynamometer. The patient will also complete the WORC questionnaire.

Surgical Technique

All patients will undergo a 15-point arthroscopic shoulder examination as per the method outlined by Snyder. An arthroscopic acromioplasty will be performed if needed according to the technique described by Snyder. The bursal side of the tear will be evaluated. If the cuff can be re-approximated to its anatomic position on the greater tuberosity without excessive tension, a standard rotator cuff reconstruction will be attempted. If this is not possible the surgeon will determine that the cuff is "irreparable" and the randomization envelope will be opened.

Wong et al. described the surgical procedure for patients in the "Bridging" group. The bursa will be debrided thoroughly and rotator cuff edges will be shaved down to stable tissue. Following this, an acellular human dermal patch will be rehydrated in saline solution for 15 minutes. The patch is stretched to remove the manufacturing surface irregularities. The patch is then sewn in place with braided polyester suture material. Multiple sutures, approximately 5 to 10 mm apart from one another will be used. The medial sutures are placed into the remnants of supraspinatus and infraspinatus tendons. The patch is then attached to the greater tuberosity in a double row configuration.

The technique described by Burkhart et al will be followed for patients in the "SCR" group. The bursa will be debrided thoroughly and rotator cuff edges will be shaved down to stable tissue. Following this, an acellular human dermal patch will be rehydrated in saline solution for 15 minutes. The patch is stretched to remove the manufacturing surface irregularities. Measurement of defect size (coronal and sagittal) will take place, following that the glenoid and humeral footprint preparation will be performed utilizing an arthroscopic burr, arthroscopic bone anchors will be inserted on the glenoid footprint and graft is inserted with double pully technique. The graft is then tensioned to greater tuberosity using a double row configuration.

Postoperative protocol

The shoulder will be immobilized in a sling for one week postoperatively, and only passive forward flexion and external rotation will be allowed for eight weeks. The patient then progresses to active shoulder motion. Strengthening will begin at twelve weeks postoperatively.

The patient will follow-up with the attending surgeon (IW) at 2 weeks post-operatively for a wound check. Then further follow-up appointments will be at 6 weeks, 3 months, 6 months, 12 and 24 months, as per current clinical practice.

At the 3, 6, 12, and 24 month visits the patient will again undergo the structured clinical examination conducted by a sports medicine fellowship trained orthopaedic consultant who is blinded to the patients' treatment group. The patient will also complete the (WORC) questionnaire at these follow-up appointments. Radiograph will be taken also to obtain the postoperative measurements. MRI will be done to assess healing at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Magnetic resonance imaging (MRI) proven diagnosis of a large or massive (>3cm), two-tendon (supraspinatus and infraspinatus) tear of the shoulder rotator cuff

Exclusion Criteria:

* Presence of subscapular tear
* Presence of glenohumeral osteoarthritis
* WORC score > 70%
* Uncontrolled diabetes
* Pregnancy
* Presence of local or systemic infection
* Paralysis of the shoulder
* Poor nutritional state
* Contracture of the shoulder
* Presence of cuff tear arthropathy
* MRI proven nonvascular surgical sites
* Cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Maintenance of Acromiohumeral Distance | 24 months
  The primary objective of this study is to compare the effect between the two surgical techniques, arthroscopic SCR for a massive, chronic irreparable tear of the rotator cuff vs. BRR with an acellular human dermal allograft implant, on the maintenance of the Acromiohumeral distance. Acromiohumeral Distance is measured in mm and determine through xray.

SECONDARY OUTCOMES:
Changes in Shoulder Strength After Surgery | 24 months
  Changes in Strength After Surgery will be measured in kilograms using a hand dynamometer.
Changes in Shoulder Range of Motion After Surgery | 24 months
  Changes in Shoulder Range of Motion After Surgery will be measured in degrees using a goniometer.
Changes in Patient Reported Outcomes using the Western Ontario Rotator Cuff Index (WORC) | 24 months
  The Western Ontario Rotator Cuff Index is a questionnaire use to evaluate patient reported outcomes. The questionnaire asks 21 questions are using a 100mm visual analogue type scale patients are asked to indicate how much pain they are experiencing doing different activities. The left end of the line indicates no pain, the right end of the line indicates extreme pain. The distance in mm from the left end of the line determines the amount of pain. To total distances for all 21 questions is added up then subtracted from 2100 and divided by 21 to give a percentage. A percentage of 100 indicates that no pain is being felt and low percentages indicates the patient is experiencing extreme pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan H Wong, MD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada